CLINICAL TRIAL: NCT04172467
Title: Quality Assurance on Diagnosis and Therapy of Secondary Immunodeficiencies (SID) in Patients With Chronic Lymphocytic Leukemia (CLL) or Multiple Myeloma (MM) in Germany (QS-SID)
Brief Title: Quality Assurance of Secondary Immunodeficiencies (SID) in CLL/MM Patients
Acronym: QS-SID
Status: Completed | Type: Observational
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Prof. Hartmut Link (Unknown); Takeda (Industry); MMF GmbH (Industry); AIO AG Supportivtherapie (Other); AG Supportive Maßnahmen in der Onkologie (Other)
Responsible Party: Sponsor
Other Study IDs: AIO-SUP-0119ass (QS SID)
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-11

CONDITIONS: Secondary Immunodeficiencies (SID)
Keywords: Secondary immunodeficiencies (SID); Chronic lymphocytic leukemia (CLL); Multiple myeloma (MM)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-interventional retrospective epidemiological observational study — non-interventional retrospective epidemiological observational study

SUMMARY:
Retrospective, representative registry for quality assurance on diagnosis and therapy of secondary immunodeficiencies (SID) in patients with chronic lymphocytic leukemia (CLL) or multiple myeloma (MM)

DETAILED DESCRIPTION:
Treatment structure analysis and recruitment (phase 1):

In a first step, data on care facilities, that treat patients with CLL or MM in Germany is obtained.

In phase 1 all centers in Germany that potentially treat patients with the CLL or MM are contacted and data of its facility care level and its number of treated patients is recorded using a one-sided pen-to-paper form. In addition, the willingness of care facilities to become involved in patients' documentation is elicited (phase 2).

Patient documentation (phase 2)

To achieve a reliable, representative sample of patients treated in Germany, the distribution of cases to be documented is specified in the individual indications amongst the facilities involved. This is done using the facilities' data on patient numbers and treatment structure obtained in phase I:

The participating centers are assigned to clusters based on key distinguishing features (facility type, care level and number of patients treated). This sample is modulated according to the previous treatment structure analysis. By taking this approach, the actual percentages of the various care facilities in an indication area can be reflected proportionally in the patient documentation sample.

In phase 2 a electronic case record form (eCRF) is completed in order to collect the original patient and treatment data, which are relevant to the purpose of the study. All data is gathered retrospectively and anonymously using the patient files. Patient and disease related variables (age, general condition according to the Eastern Cooperative Oncology Group (ECOG), relevant comorbidity, staging and relevant mutations), systemic antineoplastic treatment (chemotherapy, antibodies, kinase-inhibitors, relevant co-medication etc.) are recorded. Also, data on diagnosis of Ig-levels (IgG, IgA, IgM), therapy of secondary immunodeficiencies as well as the number and severity of occurred infections and their treatment is collected. Clusters for classification of infections will be developed (e.g. life-threatening, need for hospitalization).

In order to ensure data quality, the scientific project lead will provide training for two employees of the commissioned institute on matters regarding the content of the study. This knowledge will be incorporated into the programming of the user interface and the patient databases so that the program will check for completeness and, as far as possible, plausibility, on the basis of defined requirements and constraints. These checks accompany the process of entering data into the eCRF and allow for validating data instantly. If inconsistencies, mistakes or omissions are detected, data will be validated by an integrated query management system.

Physicians questionnaire (phase 3)

In an additional step and alongside the patient documentation, the attending physicians in participating centers will be surveyed (phase 3) on their competency profile, their assessment of guideline quality and their approach to avoid infections of CLL and MM patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with CLL or MM
* anti-neoplastic systemic therapy (all therapy lines) between July 1st 2017 and June 30th 2018

Exclusion Criteria:

- patient in terminal phase of the disease, life expectancy less than three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lymphocytic leukemia (CLL) or multiple myeloma (MM).
Sampling Method: Non-Probability Sample
Enrollment: 1086 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Link, Prof. Dr., Principal Investigator — AIO AG Supportive Therapie
Locations (1):
- Privatärztliche Praxis; Innere Medizin, Hämatologie, Internistische Onkologie, Kaiserslautern, Germany

IPD SHARING:
Plan to Share IPD: No
Data is collected retrospectively and completely anonymously from patient records, no identifying characteris-tics (e.g. birth date, initial letters, pseudonym) will be collected.
  It is hoped that these data will assist in creating new possibilities and ways to improve the quality of treatment through further training and enhancement of the availability and transparency of the guidelines.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a retrospective sample analysis of patients from practices and hospitals in Germany who were representatively screened using previously collected care parameters of the participating institutions. Previous and current treatment and infection data were collected from patients who received a line of therapy for the treatment of CLL or MM started in 2018 (1st, 2nd and 3rd or higher line).
Pre-assignment Details: The time period was chosen to ensure that patients have been followed up for at least 12 months in order to collect data on susceptibility to infection and possible secondary immunodeficiencies
Groups:
- Not Applicable. Non-interventional Retropspective Observational Study.: This was a retrospective sample analysis representative for practices and hospitals in Germany. The treatments and infection data were collected from patients with chronic lymphocytic leukaemia (CLL) and multiple myeloma (MM). GL adherence (GLAD) was analysed.
Period: Overall Study
Arm/Group | Not Applicable. Non-interventional Retropspective Observational Study.
Started | 1086
Completed | 1086
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with chronic lymphocytic leukaemia and multiple myeloma and systemic treatment in 2018
Groups:
- Non-interventional Retrospective Observational Study.: This was a retrospective sample analysis representative for practices and hospitals in Germany. The treatments and infection data were collected from patients with chronic lymphocytic leukaemia (CLL) and multiple myeloma (MM). GL adherence (GLAD) was analysed.
Arm/Group | Non-interventional Retrospective Observational Study.
Number analyzed (Participants) | 1086
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 267
  >=65 years | 819
Age, Continuous [Mean (Full Range); unit: years] — Age at the start of the therapy line under investigation
  years | 73 [33 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 475
  Male | 611
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1086
Region of Enrollment [Count of Participants; unit: Participants] — This was a retrospective sample analysis of patients from practices and hospitals in Germany who were representatively screened using previously collected care parameters of the participating institutions. Previous and current treatment and infection data were collected from patients who received a line of therapy for the treatment of CLL or MM started in 2018 (1st, 2nd and 3rd or higher line). The time period was chosen to ensure that patients have been followed up for at least 12 months in order to collect data on susceptibility to infection and possible secondary immunodeficiencies.
  Participants
    Germany | 1086
Therapy Line [Count of Participants; unit: Participants]
  1st line | 539
  2nd line | 317
  3rd line | 230
Disease [Count of Participants; unit: Participants]
  Chronic Lymphocytic Leukaemia (CLL) | 490
  Multiple Myeloma (MM) | 596

OUTCOME MEASURES:

1. Primary Outcome: Guideline Adherence (GLAD)
Description: For SID, immunoglobulin substitution (IgRT) is mandatory only for patients with an IgG level < 4g/l (or IgG subclass deficiency) and additionally more than 3 infections or a severe infection (≥ grade 3) and is optional (may be appropriate) if IgG level < 4g/l and/or 1-3 less severe infections (≤ grade 2). IgRT is not indicated if patients do not fulfil either condition.
  Scoring system:
  GLAD-Score 2: full guideline adherence GLAD-Score 1: deviations in dose or interval (+/- 10%) or a late start of IgRT (>28 days after a severe infection (≥ grade 3).
  GLAD-Score 0: IgRT without indication (overuse) or omitted IgRT despite recommendation (underuse). Likewise, 0 points were awarded if both the dose and the interval deviated from the GL recommendations (e.g. underdosed single dose) or if IgRT was not started until more than 3 months after hypogammaglobulinemia and at least one severe infection.
Time Frame: Median study observation period of 18.2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Non-interventional Retrospective Observational Study.
Number analyzed (Participants) | 1086
Participants
  GLAD-Score 2 | 889
  GLAD-Score 1 | 75
  GLAD-Score 0 | 122

2. Secondary Outcome: Guideline Adherence and Susceptibility to Infection
Description: For the analysis of susceptibility to infection, the time to next infection was examined using the Andersen-Gill model for recurrent events. For effect estimation, hazard ratios are reported with 95% confidence interval in each case. GLAD-Score 2 is Reference, a higher hazard ratio means a higher susceptibility to infection.
Time Frame: Median study observation period of 18.2 months
Measure: Number; unit: Number of infectious events
Groups:
- GLAD-Score 2: 2 points for full GLAD
- GLAD-Score 1: 1 point for deviations in dose or interval (+/- 10%) or a late start of IgRT (>28 days after a severe infection (≥ grade 3)
- GLAD-Score 0: 0 points for IgRT without indication (overuse) or omitted IgRT despite recommendation (underuse). Likewise, 0 points were awarded if both the dose and the interval deviated from the GL recommendations (e.g. underdosed single dose) or if IgRT was not started until more than 3 months after hypogammaglobulinemia and at least one severe infection
Arm/Group | GLAD-Score 2 | GLAD-Score 1 | GLAD-Score 0
Number analyzed (Participants) | 889 | 75 | 122
Number of infectious events | 250 | 63 | 221
Statistical Analysis 1: Comparison: GLAD-Score 2 vs GLAD-Score 0; For the analysis of susceptibility to infection, the time to next infection was examined using the Andersen-Gill model. This model is an extension to the proportional hazard model (Cox model) for time to recurrent event analysis. The null hypothesis is that the GLAD-Score has no effect on susceptibility to infection; Test type: Other — To estimate the relevance of guideline adherent treatment (GLAD) for the susceptibility to infection, full GLAD is taken as reference category; p < 0.001, Regression, Cox — For effect estimation, hazard ratios are reported with 95% confidence interval. The significance level is set to two-sided ≤ 5% (p ≤ 0.05); The Model developed by Anderson and Gill (1982) is an extension to the proportional hazard model (Cox model) for time to recurrent event analysis; Hazard Ratio (HR) = 4.49, 95% CI 2-sided [3.72 to 5.42]
Statistical Analysis 2: Comparison: GLAD-Score 2 vs GLAD-Score 1; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.001, Regression, Cox — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 2.52, 95% CI 2-sided [1.98 to 3.21]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Since this is an observational study of clinical routine, there is no studied medicinal product involved in this study and no safety event were extracted as part of this study.
Groups:
- Non-interventional Retropspective Observational Study.: Data from 1086 patients (CLL 490, MM 596) were collected from 86 centres.
Arm/Group | Non-interventional Retropspective Observational Study.
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The limitations of the retrospective study are that the information in the patient records cannot be verified and that the diagnosis and monitoring of the patients are not specified. In the case of infections, the classification was missing for a large number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT04172467/Prot_SAP_000.pdf